CLINICAL TRIAL: NCT04950790
Title: A Randomized, Double-blind, Placebo-parallel-controlled, Multicenter Clinical Trial of the Efficacy and Safety of Shuxinin Injection in the Treatment of Acute Ischemic Stroke
Brief Title: Study on the Effectiveness and Safety of Shuxinin Injection in the Treatment of Acute Ischemic Stroke
Status: Unknown | Phase: Phase 4 | Type: Interventional
Last Known Status: Recruiting
Sponsor: Peking University Third Hospital (Other)
Collaborators: Handan Central Hospital (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Double | Purpose: Treatment
Other Study IDs: D2018041
Record Dates: First submitted 2021-06-27; First posted 2021-07-06 (Actual); Last update posted 2021-07-07 (Actual); Status verified 2021-06

CONDITIONS: Acute Ischemic Stroke
MeSH Terms: conditions — Ischemic Stroke

STUDY DESIGN:
Who Masked: Participant, Care Provider
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Test group (Experimental): Shuxuening injection + basic treatment
  Interventions: Drug: Shuxinin injection; Drug: Basic treatment
- Control group (Placebo Comparator): placebo (sterilized water for injection) + basic treatment
  Interventions: Drug: Basic treatment; Drug: Placebo

INTERVENTIONS:
Drug: Shuxinin injection — Shuxuening injection : 5ml/ injection, intravenous infusion, 20ml each time, once a day, diluted 250ml with normal saline, 15-30 drops/min.
  Arms: Test group
Drug: Basic treatment — Give oral aspirin enteric soluble tablets 150-300mg/d as early as possible after the onset of the disease, which can be changed to a prophylactic dose (50-325mg/d) after the acute phase. For those who cannot tolerate For those who cannot tolerate aspirin, clopidogrel can be used.
Drug: Placebo — sterilized water for injection，5ml/ injection, intravenous infusion, 20ml each time, once a day, diluted 250ml with normal saline, 15-30 drops/min.
  Arms: Control group

SUMMARY:
This is a randomized, double-blind, placebo-parallel-controlled multiplier designed to observe and evaluate the efficacy and safety of Shuxuening injection in the treatment of acute ischemic stroke for 10 days and continue follow-up to 90 days after the onset of the disease.

DETAILED DESCRIPTION:
Cerebral infarction (CI), also known as ischemic stroke, refers to the softening and necrosis of local brain tissue due to blood circulation disorders, ischemia, and hypoxia. According to the 2016 Stroke Epidemiology Report [4], there are currently 70 million stroke patients in my country, 2 million new strokes occur each year, and 1.65 million deaths due to stroke each year. There is one Chinese every 12 seconds. Stroke occurs, and one Chinese person dies of a stroke every 21 seconds. Chinese people who die from a stroke each year account for 22.45% of all deaths. According to the results of the study on the incidence and mortality of stroke in the Chinese population, stroke is currently the number one cause of death in China, accounting for 20% of deaths in urban populations and 19% in rural areas. Cerebral infarction is a disease with high morbidity, high disability, high mortality and high recurrence rate in China, and it has gradually attracted widespread attention from the whole society. Shuxuening injection is developed by Shiyao Yinhu Pharmaceutical Co., Ltd., and is a sterile aqueous solution made of ginkgo biloba or ginkgo biloba extract. The auxiliary materials are ethanol and vitamin C. Its main function is to expand blood vessels and improve microcirculation. It is used for ischemic cardiovascular and cerebrovascular diseases, coronary heart disease, angina pectoris, cerebral embolism, cerebral vasospasm, etc. This trial is a randomized, double-blind, placebo-controlled multicenter clinical trial. The aim was to observe the effectiveness and safety of Shuxuening injection in the treatment of acute ischemic stroke for 10 days, and to continue follow-up to 90 days after the onset.

ELIGIBILITY:
Inclusion Criteria:

1. meeting the diagnostic criteria for acute ischemic stroke;
2. Patients with complete anterior circulation infarction (TACI), partial anterior circulation infarction (PACI), lacunar infarction (LACI) in OCSP classification;
3. Patients within 72 hours after onset;
4. NIHSS score ≥4 points and ≤17 points;
5. The modified Rankin Scale (MRS) score was between 0 and 1, and the MRS score before inclusion was > 2;
6. Aged between 40 and 80 (including 40 and 80); 7) Signing the Informed Consent.

Exclusion Criteria:

1. intracranial hemorrhagic disease indicated by head CT or MRI, or disease with bleeding tendency;
2. Patients treated with vascular opening (such as thrombolysis, arterial thrombectomy, ultra-early thrombosis aspiration and stenting, etc.) after the onset of this disease;
3. Cerebral embolism caused by brain tumor, brain injury, brain parasitic disease, metabolic disorder, rheumatic heart disease and coronary heart disease confirmed by examination;
4. Patients with other diseases affecting limb mobility, such as claudication, osteoarthritis (active stage), rheumatoid arthritis (active stage), gouty arthritis and other limb mobility disorders that may affect neurological function examination;
5. Patients with post-treatment systolic blood pressure ≥180 mmHg or fasting blood glucose concentration < 2.8mmol/L;
6. patients with severe heart and lung diseases and chronic liver and kidney dysfunction, including 1.5 times of the upper normal limit of liver function ALT and AST > and 1.2 times of the upper normal limit of renal function serum creatinine (SCR) >);
7. patients with complicated mental illness who are unable or unwilling to cooperate;
8. People with known allergies to the drug and its components (including excipients such as ethanol) and allergic constitution;
9. Any other patients considered by the investigator to be unsuitable for inclusion or to be affected by factors affecting study participation or completion;
10. Patients enrolled in other clinical trials within 1 month.

Ages: 40 Years to 80 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 480 (Estimated)
Dates: Start 2018-04-01 (Actual); Primary Completion 2021-12-01 (Estimated); Study Completion 2021-12-01 (Estimated)

PRIMARY OUTCOMES:
mRS score | baseline
  Percentage of patients with mRS score ≤2 at 90 days post-onset.
mRS score | 10 days after treatment
  Percentage of patients with mRS score ≤2 at 90 days post-onset.
mRS score | 30 days after onset
  Percentage of patients with mRS score ≤2 at 90 days post-onset.
mRS score | 90 days after onset
  Percentage of patients with mRS score ≤2 at 90 days post-onset.

CONTACTS AND LOCATIONS:
Overall Officials: Xiaogang Li, Principal Investigator — Peking University Third Hospital
Locations (1):
- Peking University Third Hospital, Beijing, China

IPD SHARING:
Plan to Share IPD: No